CLINICAL TRIAL: NCT05862103
Title: Long-Term Follow-Up in Patients With Acute Myocardial Infarction Cohort - a Prospective, Multicenter Study
Brief Title: Long-Term Follow-Up in Patients With Acute Myocardial Infarction Cohort
Status: Recruiting | Type: Observational
Sponsor: Yu Bo (Other)
Responsible Party: Sponsor-Investigator, Yu Bo, Director, Harbin Medical University
Organization: Harbin Medical University (Other)
Other Study IDs: KY2022-266
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction; Adverse Event
Keywords: Acute myocardial infarction; Major adverse cardiac and cerebrovascular event; Optimized treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- optimized group: the patients received at least one optimized treatment
  Interventions: Other: Treatment Strategies
- un-optimized group: the patients didn't receive optimized treatment

INTERVENTIONS:
Other: Treatment Strategies — AMI emergency treatment process, pre-reperfusion medication, reperfusion strategy selection, and early cardiac rehabilitation after reperfusion
  Groups: optimized group

SUMMARY:
AMI Survivors who participated in the project "Construction and key technology research of the whole myocardial protection system for acute myocardial infarction" (project number 2016YFC1301100) and completed the 1-year visit were followed up by telephone at 3 years (within the corresponding follow-up time window) and 5 years after discharge to acquire the patients' medication, health status, and major adverse cardiovascular and cerebrovascular events, including death, heart failure, rehospitalization, re-myocardial infarction, revascularization, stroke, malignant arrhythmia, and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* AMI survivors who participated in the project "Construction and key technology research of the whole myocardial protection system for acute myocardial infarction" and completed the 1-year visit.
* Telephone to obtain informed consent from the subjects/family members of the subjects.

Exclusion Criteria:

* Not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMI survivors who participated in the project "Construction and key technology research on the whole myocardial protection system for acute myocardial infarction" and completed 1-year visit
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACCE | 5 years after discharge
  the incidence of MACCE (death, heart failure, rehospitalization, re-myocardial infarction, re-myocardial revascularization, stroke, malignant arrhythmia, bleeding events, etc.) in AMI patients

SECONDARY OUTCOMES:
Differences of MACCE between the optimized group and the non-optimized group | 5 years after discharge
  Differences of the MACCE between the optimized group and the non-optimized group
Differences of the MACCE between OCT-guided group and the coronary angiography -guided group | 5 years after discharge
  Differences of the MACCE between OCT-guided group and the coronary angiography -guided group
Differences of MACCE between defer PCI group and direct PCI group | 3 and 5 years after discharge
  Differences of MACCE between defer PCI group and direct PCI group
Differences of the MACCE incidence between cardiac rehabilitation quality improvement group and non-cardiac rehabilitation group | 5 years after discharge
  Differences of the MACCE incidence between cardiac rehabilitation quality improvement group and non-cardiac rehabilitation group

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Study Chair — The Second Affiliated Hospital of Harbin Medical University
Locations (18):
- China (18):
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guangdong general hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Guangxi medical university, Nanning, Guangxi
  - Second hospital of hebei medical university, Shijiazhuang, Hebei
  - Daqing Oil Field Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The econd Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Northern Theater Command of the Chinese People's Liberation Army, Shenyang, Liaoning
  - Xijing Hospital of Air Force Military Medical University, Xi’an, Shanxi
  - Xinqiao Hospital Army Medical University, Chongqing, Sichuan
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No